CLINICAL TRIAL: NCT03888950
Title: Early Response Assessment With Interim FDG PET-CT Imaging in Patients With Advanced Melanoma Treated by Immune Checkpoint Inhibitors Therapy Anti-PD1
Brief Title: Interim FDG PET-CT in Melanoma Metastatic Patient's Treated by Anti-PD1 Therapy
Acronym: TEP-ANTI-PD1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-AOIP-02
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- early research PET-CT (Experimental): The patient will undergo an early research PET-CT after 2 cycles of anti-PD1 (PET1) between the baseline PET-CT and the PET-CT at 3 months of initiation of treatment
  Interventions: Diagnostic Test: FDG PET-CT

INTERVENTIONS:
Diagnostic Test: FDG PET-CT — FDG PET/CT for oncological imaging of adult patients

SUMMARY:
The objective of this study is to assess whether FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET-CT could be an early predictive method of therapeutic response to anti-PD-1 immunotherapy in metastatic melanoma after 2 cycles of ANTI-PD1.

20 patients will be enrolled and undergo three PET/CT scans: a baseline PET-CT, an early research PET-CT after 2 cycles of anti-PD1 (PET1) and a PET-CT at 3 months of initiation of treatment. Treatment response on FDG PET-CT will be assessed according to PERCIST criteria.

DETAILED DESCRIPTION:
The management and prognosis of patients with metastatic cutaneous melanoma have changed dramatically with the advent of immunotherapy, especially anti-PD-1 antibodies. These immune-checkpoint inhibitor block the programmend cell death receptor 1 (PD1). Currently, two anti-PD-1 antibodies, nivolumab and pembrolizumab are available. Recent data for pembrolizumab show that the overall survival rate at almost 3 years is 50% and the overall response rate is 42%. Despite these results so far never achieved, about 60% of patients do not respond to anti-PD-1 immunotherapy and, at present, no clinical, imaging or biological markers are predictive of the therapeutic response. The identification of such markers is essential in order to guide the clinician in the choice of optimal treatment.

The objective of this study is to assess whether FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET-CT could be an early predictive method of therapeutic response to anti-PD-1 immunotherapy in metastatic melanoma.

The anti-tumor immune response to anti-PD-1 is related to the activation of immune cells infiltrating the tumor, in particular CD8+ (cluster of differentiation 8) T cells whose phenotype is that of "exhausted T cells". This immune activation is such that it sometimes causes (about 10% of cases) a transient increase in the size and/or number of lesions. This phenomenon, has been called "pseudo-progression" and it cannot be interpreted routinely by RECIST1.1 criteria. The exact kinetics and timing of CD8+ T cell activation leading to response to treatment is still unknown. It is possible that this cellular activation has an early metabolic translation detectable by 18FDG PET-CT. The investigator's hypothesis is that early 18FDG PET-CT, ie after 2 cycles of anti-PD1 in metastatic patient melanoma, could be predictive of the therapeutic response. 20 patients will be enrolled and undergo three PET/CT scans: a baseline PET-CT (PET0) before the start of anti-PD1 treatment, an early PET-CT after 2 cycles of anti-PD1 (PET1) and a third PET-CT after 3 months of initiation of treatment. Treatment response on FDG PET will be assessed according to PERCIST criteria. Changes in FDG uptake will be correlated with blood results.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years,
* Patient with advanced melanoma proved histologically, not BRAF mutated, BRAFV600 mutated and wild mutated, cutaneous or unknown primary melanoma having an indication of treatment with anti-PD-1 immunotherapy by nivolumab or Pembrolizumab,
* Patient having social insurance,
* Patient who has signed informed consent.

Exclusion Criteria:

* Age less than 18 years,
* Patient with ocular or mucosal melanoma,
* Contraindication to PET CT examination: Severe claustrophobia, unbalanced diabetes (fasting hairy blood glucose ≥ 11 mmol),
* Patient with only metastatic lesions less than 8 mm in size, with the exception of pulmonary nodules,
* HIV and/or HCV (hepatitis C virus) and/or HBV (hepatitis B virus) positive serology, active autoimmune disease,
* Withdrawal of informed consent,
* Metastatic disease not confirmed histologically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quantifying changes in FDG uptake according to PERCIST criteria:Single-lesion analysis | Before the start of anti-PD1 treatment (PET0)(day 0), after 2 cycles of anti-PD1 (PET1) (between day 21 and day 31) and after 3 months of initiation of treatment(PET2)
  -Single-lesion analysis: by measuring % change in SULpeak of the one lesion with the highest SUL on PET0 and PET1 and PET2 (not necessarily the same lesion),
Quantifying changes in FDG uptake according to PERCIST criteria: Five lesion analysis | Before the start of anti-PD1 treatment (PET0)(day 0), after 2 cycles of anti-PD1 (PET1) (between day 21 and day 31) and after 3 months of initiation of treatment(PET2)
  - Five lesion analysis: by summing the SULpeak of up to 5 lesions with highest FDG uptake (maximum of two per organ).
Determine the number of lesions | Before the start of anti-PD1 treatment (PET0)(day 0), after 2 cycles of anti-PD1 (PET1) (between day 21 and day 31) and after 3 months of initiation of treatment(PET2)

SECONDARY OUTCOMES:
Analysis of SUL peak of the most avid lesions | Before the start of anti-PD1 treatment (PET0)(day 0), after 2 cycles of anti-PD1 (PET1) (between day 21 and day 31) and after 3 months of initiation of treatment(PET2)

CONTACTS AND LOCATIONS:
Overall Officials: Micheline RAZZOUK-CADET, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, CHU de NICE, France

IPD SHARING:
Plan to Share IPD: No